CLINICAL TRIAL: NCT00222404
Title: Pharmacogenomic Study Realized Within the Framework of the Common Care to "Non-small Cell Lung Carcinoma" at Any Stages Treated by Chemotherapy.
Brief Title: Pharmacogenomic Study Realized on "Non-small Cell Lung Carcinoma"
Acronym: Pharmacogenos
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: University Hospital of Grenoble, DRC
Other Study IDs: DCIC 04 40
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; Pharmacogenomic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to correlate molecular genetic profile with response to chemotherapy in case of primary chemotherapy treatment for non-small cells lung carcinoma.

DETAILED DESCRIPTION:
Lung carcinoma will be the fifth death cause in the world in 2020. In Europe it causes more deaths than carcinoma of breast, colon and prostate combined so it is a public healthcare priority. Applying high throughput molecular analysis technologies to pharmacogenomics could improve lung carcinoma care strategies. The study hypothesis is that the determination of the genomic and proteomic profiles of non-small cell lung carcinoma patients will allow treatment targeting , improving treatment efficacy and tolerance.

In order to carry out this study, the five thoracic oncology centers of the Rhône-Alpes region will collaborate with several INSERM (French national research institute) units and new biotechnology companies.

The primary objective of this study is to correlate molecular genetic profile with response to chemotherapy in cases of primary chemotherapy treatment for non-small cell lung carcinomas.

Biological samples will be collected before and during patient care to correlate clinical evolution (response and tolerance) with:

* circulating cell polymorphism profile
* proteomic profile
* genetic and epigenetic modifications of genes involved in DNA repair, drugs metabolism, apoptosis cell regulation mechanisms, and cell mobility and adhesion mechanisms.

The main judgment criteria will be response to chemotherapy correlated with patient's biological profile.

Second judgment criteria will be overall survival and hematology toxicity which will be evaluated each new cycle of chemotherapy.

The second purpose of this study is to validate less invasive methods of sampling using blood, expectoration, urine, fixed biopsies and lungs tapping, as a substitute to the current reference (frozen tumor), which is out of reach in clinical examination.

This will contribute to setting of a multicentric resources bank, to define targets for new drugs and to develop oligoarrays allowing adapted chemotherapies.

Two previous studies (1800 and 500 patients respectively) have already been carried out, data and samples are available.

For this study, 600 patients will be included over 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 suffering from Non-Small-Cell Lung Carcinoma
* Patient treated by chemotherapy with platinum salt
* Every stage TNM classification
* No previous chemotherapy
* One measurable lesion out of nervous central system at least
* Performance status from 0 to 2 on ECOG scale
* Life expectancy > 12 weeks

Exclusion Criteria:

* Previous or Concomitant carcinoma over 5 last years
* Concomitant radiotherapy
* Cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient older than 18 suffering from Non-Small-Cell Lung Carcinoma
  * Patient treated by chemotherapy with platinum salt
  * Every stage TNM classification
  * No previous chemotherapy
  * One measurable lesion out of nervous central system at least
Sampling Method: Non-Probability Sample
Enrollment: 556 (Actual)
Dates: Start 2005-07; Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chritian Brambilla, Pr., Study Director — INSERM U578
Locations (1):
- University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Beer DG, Kardia SL, Huang CC, Giordano TJ, Levin AM, Misek DE, Lin L, Chen G, Gharib TG, Thomas DG, Lizyness ML, Kuick R, Hayasaka S, Taylor JM, Iannettoni MD, Orringer MB, Hanash S. Gene-expression profiles predict survival of patients with lung adenocarcinoma. Nat Med. 2002 Aug;8(8):816-24. doi: 10.1038/nm733. Epub 2002 Jul 15. PMID 12118244
- [Background] Dumontet C, Sikic BI. Mechanisms of action of and resistance to antitubulin agents: microtubule dynamics, drug transport, and cell death. J Clin Oncol. 1999 Mar;17(3):1061-70. doi: 10.1200/JCO.1999.17.3.1061. PMID 10071301
- [Background] Dumontet C, Morschhauser F, Solal-Celigny P, Bouafia F, Bourgeois E, Thieblemont C, Leleu X, Hequet O, Salles G, Coiffier B. Gemcitabine as a single agent in the treatment of relapsed or refractory low-grade non-Hodgkin's lymphoma. Br J Haematol. 2001 Jun;113(3):772-8. doi: 10.1046/j.1365-2141.2001.02795.x. PMID 11380469
- [Background] Galmarini CM, Mackey JR, Dumontet C. Nucleoside analogues and nucleobases in cancer treatment. Lancet Oncol. 2002 Jul;3(7):415-24. doi: 10.1016/s1470-2045(02)00788-x. PMID 12142171
- [Background] Howard BA, Wang MZ, Campa MJ, Corro C, Fitzgerald MC, Patz EF Jr. Identification and validation of a potential lung cancer serum biomarker detected by matrix-assisted laser desorption/ionization-time of flight spectra analysis. Proteomics. 2003 Sep;3(9):1720-4. doi: 10.1002/pmic.200300514. PMID 12973732
- [Derived] Tissot C, Toffart AC, Villar S, Souquet PJ, Merle P, Moro-Sibilot D, Perol M, Zavadil J, Brambilla C, Olivier M, Couraud S. Circulating free DNA concentration is an independent prognostic biomarker in lung cancer. Eur Respir J. 2015 Dec;46(6):1773-80. doi: 10.1183/13993003.00676-2015. Epub 2015 Oct 22. PMID 26493785
- [Derived] Toffart AC, Moro-Sibilot D, Couraud S, Merle P, Perol M, Girard N, Souquet PJ, Mastroianni B, Ferretti GR, Romand P, Chatellain P, Vesin A, Brambilla E, Brambilla C, Timsit JF. Evaluation of RECIST in chemotherapy-treated lung cancer: the Pharmacogenoscan Study. BMC Cancer. 2014 Dec 20;14:989. doi: 10.1186/1471-2407-14-989. PMID 25527907
- [Derived] Toffart AC, Pizarro CA, Schwebel C, Sakhri L, Minet C, Duruisseaux M, Azoulay E, Moro-Sibilot D, Timsit JF. Selection criteria for intensive care unit referral of lung cancer patients: a pilot study. Eur Respir J. 2015 Feb;45(2):491-500. doi: 10.1183/09031936.00118114. Epub 2014 Oct 16. PMID 25323247